CLINICAL TRIAL: NCT02066389
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Investigate the Safety and Efficacy of ABT-494 With Background Methotrexate (MTX) in Subjects With Active Rheumatoid Arthritis (RA) Who Have Had an Inadequate Response to MTX Alone
Brief Title: A Study Investigating the Efficacy and Safety of Upadacitinib (ABT-494) Given With Methotrexate (MTX) in Adults With Rheumatoid Arthritis Who Have Had an Inadequate Response to MTX Alone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-537; 2013-003984-72 (EudraCT Number)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Musculoskeletal Disease; Arthritis; Joint Diseases; anti-inflammatory agents; antirheumatic agents
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Placebo (Placebo Comparator): Participants received placebo capsules twice daily for 12 weeks.
  Interventions: Drug: Placebo
- Upadacitinib 3 mg BID (Experimental): Participants received 3 mg upadacitinib twice daily (BID) for 12 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 6 mg BID (Experimental): Participants received 6 mg upadacitinib twice daily (BID) for 12 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 12 mg BID (Experimental): Participants received 12 mg upadacitinib twice daily (BID) for 12 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 18 mg BID (Experimental): Participants received 18 mg upadacitinib twice daily (BID) for 12 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 24 mg QD (Experimental): Participants received 24 mg upadacitinib once daily (QD) for 12 weeks.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo — Tablets for oral administration
  Arms: Placebo
Drug: Upadacitinib — Tablets for oral administration
  Other Names: ABT-494
  Arms: Upadacitinib 12 mg BID; Upadacitinib 18 mg BID; Upadacitinib 24 mg QD; Upadacitinib 3 mg BID; Upadacitinib 6 mg BID

SUMMARY:
The primary objective of the study was to compare the safety and efficacy of multiple doses of upadacitinib versus placebo in adults with moderately to severely active rheumatoid arthritis (RA) on stable background methotrexate therapy who had not shown an adequate response to methotrexate alone.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with RA based on either the 1987-revised American College of Rheumatology (ACR) classification criteria or the 2010 ACR/European League against Rheumatism (EULAR) criteria for ≥ 3 months.
2. Have active RA as defined by the following minimum disease activity criteria:

   * ≥ 6 swollen joints (based on 66 joint counts) at Screening and Baseline Visits.
   * ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits.
   * high-sensitivity C-reactive protein (hsCRP) > upper limit of normal (ULN) OR positive for both rheumatoid factor and anti-cyclic citrullinated peptide (CCP) at Screening.
3. Subjects must have been receiving oral or parenteral methotrexate therapy ≥ 3 months and on a stable prescription of 7.5 to 25 mg/week for at least 4 weeks prior to Baseline Visit. Subjects should also be on a stable dose of folic acid (or equivalent) for at least 4 weeks prior to Baseline Visit. Subjects should continue with their stable doses of methotrexate and folic acid throughout the study.
4. Except for MTX, subjects must have discontinued all oral disease-modifying anti-rheumatic drugs (DMARDs) prior to Baseline Visit as specified below or for at least five times the mean terminal elimination half-life of a drug, whichever is longer:

   * ≥ 4 weeks prior to Baseline Visit for minocycline, penicillamine, sulfasalazine, hydroxychloroquine, chloroquine, azathioprine, gold formulations, cyclophosphamide
   * ≥ 8 weeks prior to Baseline Visit for leflunomide if no elimination procedure was followed, or adhere to a washout procedure (i.e., 11 days washout with colestyramine, or 30 days washout with activated charcoal)
5. Subject has a negative tuberculosis (TB) Screening Assessment. If the subject has evidence of a latent TB infection, the subject must initiate and complete a minimum of 2 weeks (or per local guidelines, whichever is longer) of an ongoing TB prophylaxis or have documented completion of a full course of TB prophylaxis, prior to Baseline Visit.
6. Subjects can be taking non-steroidal anti-inflammatory drugs (NSAIDS), acetaminophen, oral corticosteroids (equivalent to prednisone ≤ 10 mg), or inhaled corticosteroids at a stable dose for at least 4 weeks prior to Baseline Visit for stable medical conditions and should be kept at a stable dose throughout the study. NSAIDs, acetaminophen, tramadol, codeine, hydrocodone and propoxyphene taken as needed are allowed but may not be taken 24 hours prior to any study visit. Oral and inhaled corticosteroids taken as needed are allowed but may not be taken 24 hours prior to any study visit.
7. Subjects must have discontinued high potency opiates including (but not limited to): oxycodone, oxymorphone, fentanyl, levorphanol, buprenorphine, methadone, hydromorphone, and morphine at least 4 weeks prior to Baseline Visit.

Exclusion Criteria:

1. Female who is pregnant or breastfeeding.
2. Prior exposure to Janus activated kinase (JAK) inhibitor (e.g., tofacitinib, baricitinib).
3. Prior exposure to any investigational or approved biologic RA therapy.
4. Receipt of any investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives of the drug (whichever is longer) prior to Week 0 Visit.
5. Current or expected need of other immunosuppressant medications, except methotrexate. Use of oral intake of > 10 mg prednisone/day or equivalent corticosteroid therapy (see inclusion criterion 7).
6. Subject has been treated with intra-articular or parenteral administration of corticosteroids in the preceding 8 weeks prior to the Week 0 Visit.
7. Screening laboratory values meeting the following criteria:

   * Serum aspartate transaminase (AST) or alanine transaminase (ALT) > 1.5 × ULN
   * Estimated glomerular filtration rate (eGRF) by simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula < 40 mL/min/1.73 m²
   * Total white blood cell count (WBC) < 3,000/µL
   * Absolute neutrophil count (ANC) < 1,200/µL
   * Platelet count < 100,000/µL
   * Absolute lymphocytes count < 750/ µL
   * Hemoglobin < 9 gm/dL

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2015-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (63):
- United States (12):
  - C.V. Mehta MD, Med Corporation /ID# 126380, Hemet, California
  - Omega Research Consultants, LLC /ID# 125780, DeBary, Florida
  - Lovelace Scientific Resources /ID# 127324, Venice, Florida
  - North Georgia Rheumatology Grp /ID# 125779, Lawrenceville, Georgia
  - PRN Professional Research Network of Kansas, LLC /ID# 126148, Wichita, Kansas
  - The Center for Rheumatology & /ID# 127323, Wheaton, Maryland
  - Summit Medical Group /ID# 125776, Clifton, New Jersey
  - Arthritis and Osteo Assoc /ID# 134994, Las Cruces, New Mexico
  - Altoona Ctr Clinical Res /ID# 125777, Duncansville, Pennsylvania
  - Emkey Arthritis and Osteo Clin /ID# 134716, Wyomissing, Pennsylvania
  - Accurate Clinical Research /ID# 126535, Houston, Texas
  - Mountain State Clinical Resear /ID# 127089, Clarksburg, West Virginia
- Bulgaria (7):
  - MHAT Trimontsium /ID# 127311, Plovdiv
  - UMHAT Pulmed OOD /ID# 127307, Plovdiv
  - MHAT Kaspela /ID# 127315, Plovdiv
  - Diagnostic Consultative Center /ID# 127313, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 127314, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 131608, Sofia
  - Diagnostic Consultative Center /ID# 127312, Varna
- Chile (2):
  - Corp de Beneficencia Osorno /ID# 127337, Osorno
  - Quantum Research LTDA. /ID# 127338, Puerto Varas
- Czechia (4):
  - Revmatologicky ustav Praha /ID# 127317, Prague, Praha 2
  - Nuselská poliklinika, Revmatologie /ID# 127318, Prague, Praha 4
  - Revmatologie Bruntal, s.r.o /ID# 126881, Bruntál
  - Artroscan s.r.o. /ID# 126845, Ostrava
- Hungary (2):
  - Qualiclinic Kft. /ID# 127340, Budapest III, Pest County
  - Veszprem Megyei Csolnoky Feren /ID# 126876, Veszprém
- Israel (3):
  - Barzilai Medical Center /ID# 126875, Ashkelon
  - Rambam Health Care Campus /ID# 127341, Haifa
  - Sheba Medical Center /ID# 126878, Ramat Gan
- Latvia (3):
  - LTD M&M Centers /ID# 127346, Ādaži
  - Arija's Ancane's Family Doctor /ID# 127342, Baldone
  - Clinic ORTO /ID# 127345, Riga
- Mexico (3):
  - Hospital de Jesús Nazareno /ID# 127352, Mexico City
  - Cliditer SA de CV /ID# 127347, Mexico City
  - Clinstile, S.A. de C.V. /ID# 127350, Mexico City
- Poland (7):
  - Centrum Medyczne Pratia Krakow /ID# 127358, Krakow, Lesser Poland Voivodeship
  - REUMED Sp.z o.o. Filia nr 1 /ID# 127353, Lublin, Lublin Voivodeship
  - NBR Polska /ID# 127359, Warsaw, Masovian Voivodeship
  - Medica Pro Familia S.A Warszawa /ID# 127361, Warsaw, Masovian Voivodeship
  - Gabinet Internistyczno Reum. /ID# 127357, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 127360, Gdynia, Pomeranian Voivodeship
  - Michal Bazela Higher-Med /ID# 127355, Elblag, Warmian-Masurian Voivodeship
- GCM Medical Group /ID# 127363, San Juan, Puerto Rico
- Russia (3):
  - City Clinical Hospital #7 /ID# 127372, Kazan', Tatarstan, Respublika
  - Tver Regional Clinical Hosp. /ID# 127375, Tver', Tver Oblast
  - II Dzhan Research Center /ID# 127376, Saint Petersburg
- Slovakia (2):
  - MEDMAN s.r.o. /ID# 127381, Martin
  - Poliklinika Senica /ID# 127396, Senica
- South Africa (2):
  - Panorama Medical Centre /ID# 126846, Cape Town, Western Cape
  - Winelands Medical Research Ctr /ID# 126844, Stellenbosch, Western Cape
- Spain (8):
  - Hospital Regional de Malaga /ID# 127385, Málaga, Malaga
  - Hospital Plató /ID# 127384, Barcelona
  - Hospital CIMA Sanitas /ID# 127383, Barcelona
  - Hospital Universitario Basurto /ID# 127391, Bilbao
  - Hospital Clin Univ San Carlos /ID# 127382, Madrid
  - Clinica Gaias /ID# 127386, Santiago de Compostela
  - Hospital Infanta Luisa /ID# 127389, Seville
  - Hospital Universitario de Valm /ID# 127387, Seville
- Medeniyet Univ. Goztepe Traini /ID# 132396, Istanbul, Turkey (Türkiye)
- Ukraine (3):
  - Kiev Municipal Clin Hosp 3 /ID# 127419, Kiev
  - NSC-Strazhesko Ist Cardiology /ID# 127416, Kiev
  - Sumy State University /ID# 127418, Sumy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Genovese MC, Smolen JS, Weinblatt ME, Burmester GR, Meerwein S, Camp HS, Wang L, Othman AA, Khan N, Pangan AL, Jungerwirth S. Efficacy and Safety of ABT-494, a Selective JAK-1 Inhibitor, in a Phase IIb Study in Patients With Rheumatoid Arthritis and an Inadequate Response to Methotrexate. Arthritis Rheumatol. 2016 Dec;68(12):2857-2866. doi: 10.1002/art.39808. PMID 27390150
- [Derived] Yamaoka K, Tanaka Y, Kameda H, Khan N, Sasaki N, Harigai M, Song Y, Zhang Y, Takeuchi T. The Safety Profile of Upadacitinib in Patients with Rheumatoid Arthritis in Japan. Drug Saf. 2021 Jun;44(6):711-722. doi: 10.1007/s40264-021-01067-x. Epub 2021 May 27. PMID 34041702
- [Derived] Nader A, Mohamed MF, Winzenborg I, Doelger E, Noertersheuser P, Pangan AL, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy and Safety in Phase II and III Studies to Support Benefit-Risk Assessment in Rheumatoid Arthritis. Clin Pharmacol Ther. 2020 Apr;107(4):994-1003. doi: 10.1002/cpt.1671. Epub 2019 Nov 30. PMID 31610021
- [Derived] Mohamed MF, Klunder B, Camp HS, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy in Phase II Trials in Rheumatoid Arthritis and Basis for Phase III Dose Selection. Clin Pharmacol Ther. 2019 Dec;106(6):1319-1327. doi: 10.1002/cpt.1543. Epub 2019 Aug 23. PMID 31194885
- [Derived] Klunder B, Mohamed MF, Othman AA. Population Pharmacokinetics of Upadacitinib in Healthy Subjects and Subjects with Rheumatoid Arthritis: Analyses of Phase I and II Clinical Trials. Clin Pharmacokinet. 2018 Aug;57(8):977-988. doi: 10.1007/s40262-017-0605-6. PMID 29076110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 300 adults with rheumatoid arthritis (RA) were enrolled at 59 study sites located in 16 countries.
Pre-assignment Details: Eligible participants were randomly assigned in a 1:1:1:1:1:1 ratio to receive 1 of 5 doses of upadacitinib or placebo for 12 weeks.
  Participants who completed the 12-week treatment period completed a 30-day follow-up visit or had the option to enter an open-label extension study M13-538 (NCT02049138).
Period: Overall Study
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
Started | 50 | 50 | 50 | 50 | 50 | 50
Received Study Drug | 50 | 50 | 50 | 50 | 50 | 49
Completed | 45 | 49 | 44 | 47 | 43 | 45
Not Completed | 5 | 1 | 6 | 3 | 7 | 5
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 5 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 5 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Randomized in Error | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD | Total
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 49 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.51) | 53.1 (12.15) | 54.8 (12.47) | 55.7 (11.65) | 54.6 (13.65) | 56.2 (11.79) | 54.8 (12.16)
Age, Customized [Count of Participants; unit: Participants]
  18 to < 45 years | 9 | 11 | 9 | 7 | 13 | 7 | 56
  45 to < 65 years | 32 | 30 | 30 | 32 | 25 | 27 | 176
  ≤ 65 years | 9 | 9 | 11 | 11 | 12 | 15 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 34 | 41 | 42 | 42 | 237
  Male | 12 | 10 | 16 | 9 | 8 | 7 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 17 | 17 | 7 | 8 | 68
  Not Hispanic or Latino | 39 | 42 | 33 | 33 | 43 | 41 | 231
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 48 | 49 | 48 | 49 | 49 | 293
  Black or African American | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Multi-race | 0 | 1 | 0 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: All randomized participants who received at least 1 dose of study drug; last observation carried forward (LOCF) imputation was used for participants with missing data at Week 12 if prior post-baseline data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
Number analyzed (Participants) | 46 | 48 | 49 | 49 | 47 | 49
percentage of participants | 50.0 | 64.6 | 73.5 | 81.6 | 76.6 | 81.6
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 3 mg BID; Test type: Superiority; p = 0.153, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 6 mg BID; Test type: Superiority; p = 0.018, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 12 mg BID; Test type: Superiority; p = 0.001, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 18 mg BID; Test type: Superiority; p = 0.008, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 24 mg QD; Test type: Superiority; p = 0.001, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05

2. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: A participant was a responder if the following 3 criteria for improvement from baseline were met:
  * ≥ 50% improvement in 68-tender joint count;
  * ≥ 50% improvement in 66-swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Physician's global assessment of disease activity
    * Patient's global assessment of disease activity
    * Patient's assessment of pain
    * Health Assessment Questionnaire - Disability Index (HAQ-DI)
    * High sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
Number analyzed (Participants) | 46 | 48 | 49 | 50 | 47 | 48
percentage of participants | 19.6 | 39.6 | 49.0 | 50.0 | 44.7 | 43.8
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 3 mg BID; Test type: Superiority; p = 0.034, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 6 mg BID; Test type: Superiority; p = 0.003, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 12 mg BID; Test type: Superiority; p = 0.002, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 18 mg BID; Test type: Superiority; p = 0.010, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 24 mg QD; Test type: Superiority; p = 0.012, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05

3. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: A participant was a responder if the following 3 criteria for improvement from baseline were met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Physician global assessment of disease activity
    * Patient global assessment of disease activity
    * Patient assessment of pain
    * Health Assessment Questionnaire - Disability Index (HAQ-DI)
    * High sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
Number analyzed (Participants) | 46 | 47 | 49 | 50 | 47 | 48
percentage of participants | 6.5 | 23.4 | 30.6 | 16.0 | 27.7 | 25.0
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 3 mg BID; Test type: Superiority; p = 0.023, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 6 mg BID; Test type: Superiority; p = 0.003, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 12 mg BID; Test type: Superiority; p = 0.145, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 18 mg BID; Test type: Superiority; p = 0.007, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 24 mg QD; Test type: Superiority; p = 0.014, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05

4. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 12
Description: The disease activity score-28-CRP (DAS28 [CRP]) assesses RA disease activity based on a continuous scale of combined measures of 28 tender joint counts (TJC28), 28 swollen joint counts (SJC28), C-reactive protein (CRP), and the patient global assessment of disease activity (measured on a visual analog scale (VAS) from 0 to 100 mm). DAS28(CRP) scores range from 0 to approximately 10 where higher scores indicate more disease activity.
  LDA is defined as a DAS28(CRP) score < 3.2.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
Number analyzed (Participants) | 47 | 49 | 49 | 50 | 49 | 49
percentage of participants | 21.3 | 49.0 | 57.1 | 46.0 | 51.0 | 42.9
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 3 mg BID; Test type: Superiority; p = 0.005, Fisher Exact — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 6 mg BID; Test type: Superiority; p < 0.001, Fisher Exact — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 12 mg BID; Test type: Superiority; p = 0.010, Fisher Exact — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 18 mg BID; Test type: Superiority; p = 0.002, Fisher Exact — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 24 mg QD; Test type: Superiority; p = 0.024, Fisher Exact — Statistical tests were 1-sided at a significance level of 0.05

5. Secondary Outcome: Secondary: Percentage of Participants Achieving Clinical Remission (CR) Based on DAS28(CRP) at Week 12
Description: The disease activity score-28-CRP (DAS28 [CRP]) assesses RA disease activity based on a continuous scale of combined measures of 28 tender joint counts (TJC28), 28 swollen joint counts (SJC28), C-reactive protein (CRP), and the patient global assessment of disease activity (measured on a visual analog scale from 0 to 100 mm). DAS28(CRP) scores range from 0 to 10 where higher scores indicate more disease activity.
  CR is defined as a DAS28(CRP) score < 2.6.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
Number analyzed (Participants) | 47 | 49 | 49 | 50 | 49 | 49
percentage of participants | 14.9 | 36.7 | 38.8 | 34.0 | 42.9 | 22.4
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 3 mg BID; Test type: Superiority; p = 0.015, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 6 mg BID; Test type: Superiority; p = 0.008, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 12 mg BID; Test type: Superiority; p = 0.029, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 18 mg BID; Test type: Superiority; p = 0.003, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 24 mg QD; Test type: Superiority; p = 0.343, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05

6. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on CDAI at Week 12
Description: The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of TJC28 and SJC28, patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity.
  LDA is defined as a CDAI score ≤ 10.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
Number analyzed (Participants) | 47 | 49 | 49 | 50 | 49 | 49
percentage of participants | 21.3 | 40.8 | 40.8 | 40.0 | 49.0 | 36.7
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 3 mg BID; Test type: Superiority; p = 0.039, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 6 mg BID; Test type: Superiority; p = 0.039, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 12 mg BID; Test type: Superiority; p = 0.046, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 18 mg BID; Test type: Superiority; p = 0.005, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 24 mg QD; Test type: Superiority; p = 0.096, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05

7. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Based on CDAI at Week 12
Description: The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of TJC28 and SJC28, patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity.
  CR is defined as a CDAI score ≤ 2.8.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
Number analyzed (Participants) | 47 | 49 | 49 | 50 | 49 | 49
percentage of participants | 4.3 | 12.2 | 14.3 | 6.0 | 14.3 | 6.1
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 3 mg BID; Test type: Superiority; p = 0.269, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 6 mg BID; Test type: Superiority; p = 0.160, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 12 mg BID; Test type: Superiority; p = 1.000, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 18 mg BID; Test type: Superiority; p = 0.160, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 24 mg QD; Test type: Superiority; p = 1.000, Chi-squared — Statistical tests were 1-sided at a significance level of 0.05

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 30 days after last dose (up to 16 weeks).
Arm/Group | Placebo | Upadacitinib 3 mg BID | Upadacitinib 6 mg BID | Upadacitinib 12 mg BID | Upadacitinib 18 mg BID | Upadacitinib 24 mg QD
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50 | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 2/50 | 1/50 | 3/50 | 2/49
Other Adverse Events (participants affected / at risk) | 2/50 | 5/50 | 7/50 | 17/50 | 6/50 | 6/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Upadacitinib 3 mg BID (N=50) | Upadacitinib 6 mg BID (N=50) | Upadacitinib 12 mg BID (N=50) | Upadacitinib 18 mg BID (N=50) | Upadacitinib 24 mg QD (N=49)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Upadacitinib 3 mg BID (N=50) | Upadacitinib 6 mg BID (N=50) | Upadacitinib 12 mg BID (N=50) | Upadacitinib 18 mg BID (N=50) | Upadacitinib 24 mg QD (N=49)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 3 (3)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 1 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.